CLINICAL TRIAL: NCT05710679
Title: Prediction of Residual Disease by Circulating DNA Detection After Potentiated Radiotherapy for Locally Advanced Head and Neck Cancer
Acronym: NeckTAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Collaborators: GIRCI Auvergne Rhône-Alpes (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A01668-35
Record Dates: First submitted 2023-01-13; First posted 2023-02-02 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Head and Neck Carcinoma
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Biological samples of patients included in the study (i.e., patients treated with radiochemotherapy for a locally advanced head and neck cancer) will be analysed (Next generation sequencing (NGS)):
  * At inclusion : a FFPE block + a blood sample to identify tumor specific variants (tcDNA and cvDNA)
  * 3 months after radiotherapy in case of incomplete response (PET-CT) : a blood sample to search if the tumor specific variants identified before the treatment are found
  Patients with incomplete response after 3 months radiochemotherapy will undergone a salvage adenectomy.
  The main objective is to assess the ability of circulating DNA to predict residual disease during salvage adenectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional (Experimental)
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — The intervention consist in a blood sample that will be taken twice :
  * at the inclusion (before treatment)
  * 3 months after the radiochemotherapy in case of incomplete response (PET-CT)

SUMMARY:
Sixty percent of newly diagnosed head and neck squamous cell carcinomas (HNSCCs) are at a locally advanced (LA) stage. Depending on tumor site, stage, and resectability, locoregional failure rates can range from 35% to 65%. The persistence of residual disease at the end of treatment is a major prognostic element but is not always reliably assessed by current imaging techniques. Up to 40-50% of patients have residual adenomegaly and only 30% have viable disease when further adenectomy is performed. Sensitive and reproducible detection of residual disease after treatment is a major challenge in this patient category.

18F-fluorodeoxyglucose (18F-FDG) positron emission tomography-computed tomography (PET/CT) guided surveillance, with a negative predictive value of 95-97%, has proven to be non-inferior to cervical curage in HNSCCs with residual adenomegaly. Cervical curage is now indicated only if the response assessed by PET-CT is incomplete. Nevertheless, the ability of PET-CT to predict treatment failure is unsatisfactory due to a high frequency of false positives, because of inflammatory changes, with a positive predictive value of about 20-50%.

Circulating tumor DNA (ctDNA) may provide a more reliable assessment of response to potentiated radiotherapy. Liquid biopsy monitoring of response in patients treated with potentiated radiation therapy for locally advanced HNSCCs a has been shown to be feasible. In 85% of patients, ctDNA is detectable and correlates significantly with tumor volume and response to treatment. In addition, one study showed that post-radiotherapy analysis of circulating HPV16 viral DNA (cvDNA) in patients with HPV16-related HNSCCs complemented PET-CT and helped guide management decisions. HPV16 cvDNA and PET-CT have similar negative predictive values, whereas the positive predictive value is higher for HPV16 cvDNA (100% versus 50%). Nevertheless, current data are insufficient to allow routine use of this marker.

This is a multicenter, single arm, open study for patients with a locally advanced head and neck cancer for which a potentiated radiotherapy is indicated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 80 years
* Histologically confirmed, never treated squamous cell carcinoma with lymph node involvement
* squamous cell carcinoma p16+or p16-, stage III (N1), IVa or IVb (UICC classification 8th edition), N1 minimum, and oropharyngeal sqamous cell carcinomas p16+ stage I or II, N1 minimum, resectable but not operated or unresectable, with indication for concomitant or sequential radiochemotherapy with induction chemotherapy using Docetaxel, Platinum, 5-Fluorouracil (TPF or modified TPF according to the practices of the investigating centers)
* Oral cavity, oropharynx, hypopharynx or larynx, cervical adenopathies without primary
* Availability of FFPE samples prior to treatment initiation
* Detection of circulating DNA in the initial blood sample
* Obtaining informed consent from the patient
* Affiliation to the French social security system

Exclusion Criteria:

* Tumor of the nasopharynx, sinuses, nasal cavity, salivary glands or thyroid cancer
* Treatment by exclusive radiotherapy
* Contraindication to cervical lymph node dissection
* Metastatic disease (stage IVc)
* Previous treatment for head and neck cancer
* History of other cancer in the last 3 years (except carcinoma in situ, basal cell skin carcinoma, localized prostate cancer Gleason 6)
* Pregnant or breastfeeding woman
* Patient under guardianship or curators
* Psychological disorder (cognitive disorders, vigilance disorders, etc.) or social reasons (deprivation of liberty by judicial or administrative decision) or geographical reasons that could compromise the medical follow-up of the trial or compliance with the treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with incomplete cervical lymph node response on PET-CT after radiochemotherapy having circulating DNA (cDNA) | 3 months after potentiated radiotherapy
  Presence/absence of circulating DNA after treatment versus presence/absence of residual disease

SECONDARY OUTCOMES:
cDNA detection rate among patients with residual adenomegaly after treatment | at three-months after potentiated radiotherapy.
  The detection of cDNA and response on CT-Scan will be compared
Assessment of the prognostic value of cDNA detection 3 months after the end of radiochemotherapy for patients with residual adenomegaly | at three-months after potentiated radiotherapy.
  Evaluated by overall and progression-free survival
Assessment of the prognosis value of the presence of residual adenomegaly | At month 27
  Evaluated by overall and progression-free survival
Rate of concordance of mutational profiles and Human papillomavirus-high risk (HPV-HR) genotypes between the primary tumor and cDNAs at diagnosis | Inclusion
  evaluated the mutational profiles from FFPE block and the inclusion blood sample
Rate of concordance between p16 immunohistochemistry and HPV-HR genotyping on the primary tumor | Inclusion
Test of the concordance between real-time polymerase chain reaction (PCR) and NGS on formalin-fixed paraffin-embedded (FFPE) for simultaneous detection and genotyping of HPV-HR at diagnosis | Inclusion
Number of patients with ctDNA and cvDNA detection at diagnosis and the clinical, paraclinical and pathological features of the cancer | Through study completion, an average of 66 months
Evaluation of interobserver reproducibility of the interpretation of SUVmax measurements of residual cervical adenomegaly. | 3 months after potentiated radiotherapy
  A centralized review of the PET-CT will be done by the sponsor to evaluate the reproducibility of the interpretation of SUVmax measurements of residual cervixal adenomegaly (pathological/benign/equivocal)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen BERNADACH, MD, Principal Investigator — Centre Jean Perrin
Locations (3):
- France (3):
  - Centre Jean PERRIN, Clermont-Ferrand, Puy-de-Dôme
  - Hôpital de la Croix-Rousse, Lyon
  - CHU de Saint-Étienne, Saint-Etienne

REFERENCES:
- [Background] Ginzac A, Ferreira MC, Cayre A, Bouvet C, Biau J, Molnar I, Saroul N, Pham-Dang N, Durando X, Bernadach M. Prediction of residual disease using circulating DNA detection after potentiated radiotherapy for locally advanced head and neck cancer (NeckTAR): a study protocol for a prospective, multicentre trial. BMC Cancer. 2023 Jul 4;23(1):621. doi: 10.1186/s12885-023-11136-2. PMID 37400806